CLINICAL TRIAL: NCT04968977
Title: Long-term Outcomes Following Percutaneous Coronary Intervention Versus Coronary Artery Bypass Grafting for Treating In-stent Restenosis in Unprotected Left Main Coronary Artery: Multicenter LM-DRAGON Registry
Brief Title: PCI vs. CABG in UPLM-ISR
Acronym: LM-DRAGON
Status: Completed | Type: Observational
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Wojciech Wańha, MD, PhD, Medical University of Silesia
Other Study IDs: 05
Record Dates: First submitted 2021-07-09; First posted 2021-07-20 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Restenosis, Coronary; Left Main Coronary Artery Disease; PTCA Left Main Artery Complications
Keywords: unprotected left main; in-stent restenosis; coronary artery bypass graft; percutaneous coronary intervention
MeSH Terms: conditions — Coronary Restenosis; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- UPLM-ISR
  Interventions: Procedure: PCI vs. CABG

INTERVENTIONS:
Procedure: PCI vs. CABG — PCI vs. CABG

SUMMARY:
Left main (LM) coronary artery disease is associated with high morbidity and mortality owing to the large myocardial territory at risk for ischemia. Evidence from randomized controlled trials supports that percutaneous coronary intervention (PCI) with drug-eluting stents (DES) for LM disease is an acceptable treatment strategy compared with coronary artery bypass graft surgery in patients with low or intermediate anatomic complexity. However in-stent restenosis (ISR) after DES in LM disease is still occurring with an incidence of 9,7%. Studies comparing the percutaneous coronary intervention with coronary artery bypass grafting (CABG) in the treatment of in-stent restenosis in unprotected left main have been scarce. While surgical revascularization is considered to be the standard treatment for this kind of stent failure, owing to a high risk of perioperative morbidity and mortality, the restoration of flow with PCI may be a reliable alternative. Additionally, it is not clear whether re-PCI is safe in these patients. Therefore, the purpose of the present study was to compare long-term outcomes following PCI or CABG for UPLM-ISR disease.

ELIGIBILITY:
Patients were divided into two separate cohorts for the analyses. The data included consecutive patients with ≥50% diameter UPLM-ISR, with or without multivessel coronary artery disease. Patients with an equivalent of UPLM-ISR: left main distal bifurcation disease, within the proximal 5 mm of the left anterior descending artery (LAD) or left circumflex artery (LCx) ostium (in the absence of significant angiographic stenosis in the left main coronary artery), were eligible. Patients who had protected LM-ISR, defined as the occurrence of at least one patent arterial or venous graft to the left coronary artery, other concomitant non-CABG procedure during surgery, were excluded.

Age Groups: Child, Adult, Older Adult
Study Population: A total of 305 unselected patients were included in the pooled analysis, of whom 203 (66.6%) patients were treated with a PCI and 102 (33.4%) with a CABG.
Sampling Method: Probability Sample
Enrollment: 305 (Actual)
Dates: Start 2001-01-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
MACCE | 4 years

SECONDARY OUTCOMES:
cardiac death | 4 years
myocardial infarction | 4 years
target vessel revascularization | 4 years
stroke | 4 years

CONTACTS AND LOCATIONS:
Locations (11):
- Fabrizio D'Ascenzo, Turin, Italy
- Poland (10):
  - Department of Invasive Cardiology, Medical University of Bialystok, The Medical University of Bialystok Clinical Hospital, Bialystok
  - First Department of Cardiology, Medical University of Gdansk, Gdansk, Poland, Gdansk
  - Department of Cardiology and Structural Heart Diseases, Medical University of Silesia, Katowice, Poland, Katowice
  - Jacek Legutko, Krakow
  - Second Department of Cardiology, Jagiellonian University Medical College, Krakow, Poland, Krakow
  - Miedziowe Centrum Zdrowia S.A., Lubin
  - Marek Grygier, Poznan
  - Department of Invasive Cardiology, Centre of Postgraduate Medical Education, Central Clinical Hospital of the Ministry of Interior and Administration, Warsaw
  - Centre for Heart Disease, University Hospital Wroclaw Department of Heart Disease, Wroclaw Medical University, Wroclaw
  - Third Department of Cardiology, Medical University of Katowice, Zabrze

IPD SHARING:
Plan to Share IPD: Undecided
The data that support the findings of this study are available from the corresponding author upon reasonable request.

REFERENCES:
- [Derived] Wanha W, Bil J, Kolodziejczak M, Kowalowka A, Kowalewski M, Hudziak D, Gocol R, Januszek R, Figatowski T, Milewski M, Tomasiewicz B, Kubler P, Hrymniak B, Desperak P, Kuzma L, Milewski K, Gora B, Los A, Kulczycki J, Wlodarczak A, Skorupski W, Grygier M, Lesiak M, D'Ascenzo F, Andres M, Kleczynski P, Litwinowicz R, Borin A, Smolka G, Reczuch K, Gruchala M, Gil RJ, Jaguszewski M, Bartus K, Suwalski P, Dobrzycki S, Dudek D, Bartus S, Ga Sior M, Ochala A, Lansky AJ, Deja M, Legutko J, Kedhi E, Wojakowski W. Percutaneous Coronary Intervention vs. Coronary Artery Bypass Grafting for Treating In-Stent Restenosis in Unprotected-Left Main: LM-DRAGON-Registry. Front Cardiovasc Med. 2022 Apr 29;9:849971. doi: 10.3389/fcvm.2022.849971. eCollection 2022. PMID 35615559